CLINICAL TRIAL: NCT04027218
Title: Cross-over Clinical Trial to Assess the Effectiveness of Applying Dry Local Heat and/ or High Tourniquet Pressure With Current Clinical Practice for Venipuncture, and Blinded for Evaluating Their Impact on Hemolysis
Brief Title: Clinical Trial to Assess the Effectiveness of Applying Dry Local Heat and/ or High Tourniquet Pressure for Venipuncture.
Acronym: ECYPVEN-H/17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3113
Record Dates: First submitted 2019-07-12; First posted 2019-07-19 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-07

CONDITIONS: Venipuncture; Healthy Adult
Keywords: venipuncture; hemolysis; heat; pressure; safety
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Intervention Model Description: Experimental, randomized and controlled study with the usual technique of inserting a venipuncture catheter until now. Incomplete clinical trial, blind to third parties, in healthy volunteers, which consists of three arms, in which they are intervened and the comparator is applied.
Who Masked: Investigator
Masking Description: For hemolysis analysis in blood samples, the responsible of analysis by spectrophotometry is blinded from the intervention or comparator used for blood sample performed, using two different departments: one for interventions and comparator applications and other for spectrophotometer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Current clinical practice-Dry heat (Active Comparator): The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  1 period (current clinical practice) and 2 period (dry heat) or 1 period (dry heat) and 2 period (current clinical practice).
  Interventions: Device: Dry heat
- Current clinical practice- Hihg pressure (Active Comparator): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  1 period (current clinical practice) and 2 period (high pressure) or 1 period (high pressure) and 2 period (current clinical practice).
  Interventions: Device: High pressure
- Current clinical practice-Combination (Active Comparator): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  1 period (current clinical practice) and 2 period (combination of dry heat and high pressure) or 1 period (combination of dry heat and high pressure) and 2 period (current clinical practice).
  Interventions: Device: Combination of dry heat and high pressure

INTERVENTIONS:
Device: Dry heat — The application is made with two sacks of carob seeds during 7 minutes. The sacks are placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power.
  Arms: Current clinical practice-Dry heat
Device: High pressure — It will be carried out with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand (QUIRUMED) with European Conformity (CE) marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
  Arms: Current clinical practice- Hihg pressure
Device: Combination of dry heat and high pressure — The application is made with two sacks of carob seeds during 7 minutes. The sacks may be placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power; according to instructions for use.
  After 7 minutes, the pressure is applied with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand QUIRUMED with CE Marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
  Arms: Current clinical practice-Combination

SUMMARY:
Low level intervention health products clinical trial, fourth phase, non-commercial research. Dissertation of COMPLUTENSE UNIVERSITY of Madrid.

Principal Investigator of this clinical trial: Ms. LETICIA CARMEN SIMÓN LÓPEZ Collaborative investigators: Dr. DOLORES OCHOA-MAZARRO (principal investigator of bioequivalence clinical trial), and Sir. SERGIO LUQUERO-BUENO (collaborative researcher)

The setting is Clinical trials Unit of Clinical Pharmacology Department. LA PRINCESA HOSPITAL of Madrid. Research Ethical Committee of LA PRINCESA HOSPITAL of Madrid. Any person will monitor this clinical trial because the sponsor and principal researcher are the same person. Nevertheless, an adherence to this protocol will ensure by principal researcher and co-researchers.

The three interventions are:

1. To Apply local dry heat.
2. To apply high tourniquet pressure.
3. To apply both of them. (Dry heat and high pressure) The common comparator: Current Clinical practice for peripheral venous catheterization.

The main hypothesis: The number of attempts of success venipuncture at first time are influenced by any of the interventions applied before.

The main goal: To identify the most effective intervention of applying dry local heat and/or high tourniquet pressure in relation of number success venipuncture attempts, compared to current clinical practice.

Design: An experimental, randomized study which is controlled with current clinical practice to insert a peripheral vein catheter. It is an incomplete cross-over clinical trial, with three arms which are involved interventions and a common comparator.

Population: Adult healthy subjects. Sample size: It is required to enroll 54 subjects with a 95% of level of confidence and 80% level of power.

Main variable: Succeed peripheral vein catheter insertion at first attempt.

Effectiveness assessment: The optimal effectiveness is considered when vein cannulation success at first attempt exceeds 95% applying any of the interventions.

Planned date to address: It is planned to carry out around June and/or July of 2017 for the main variable.

DETAILED DESCRIPTION:
The study is considered a low level intervention clinical trial to evaluate the use and safety of a sanitary product marketed and accredited for a different aim, but according to their rules of using.

It is experimental, randomized and controlled study with the usual technique of inserting a venipuncture catheter until now. Incomplete clinical trial, blind to third parties, in healthy volunteers, which consists of three arms, in which they are intervened and the comparator is applied. The volunteers comes from a bioequivalence clinical trial for testing a new drug, and a venous catheter is required in two period between a wash-out period of one week, approximately.

For each volunteer one of intervention is applied in one period, and in other period the comparator is applied. Thus, one intervention and the sequence of one intervention application and comparator is assigned by randomization using sealed envelopes. Randomization is only performed in first period, in second period one intervention or comparator assigned in applied. Thus, each one volunteer is her/his own comparator

. Before assigned intervention or comparator is applied, a Venous International Assessment is carried out using Venous International Assessment (VIA) validated scale by nurse perception and palpation. After assigned intervention, another VIA is performed. Then, when peripheral venous catheterization is achieved, a blood sample is withdrawn in order to examine hemolysis. Afterwards, pain is registered by Visual Analogue Scale (VAS) validated scale within no more than two hours from vein catheterization, and skin perception is evaluated by Fitzpatrick's scale (only in first period) in order to analyze a possible relationship with adverse events on skin. Subjects are followed-up for 72h in order to monitor adverse events if applicable.

According to hemolysis, an ethylene diamine tetra acetate (EDTA) blood sample is processing at 3400 revolutions per minute at 4 Celsius grades for 10 minutes, and plasma samples are frosted for 24-48h. Afterwards, they are defrosted, and analyzed by absorbance using NANODROP SPECTROPHOTOMETER. The analysis by spectrophotometer is blinded of intervention or comparator used to withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form for bioequivalence study
* Signed the informed consent form for this clinical trial
* Fluid intake of participants was limited to a volume equal to or less than 500 ml
* Participants fasted 6-8 hours before venous cannulation
* Body mass index (BMI) between 18.5-29.9
* Vein perception by Venous International Assessment (VIA) scale between 5 to 2 grade.

Exclusion Criteria:

* Grade one in VIA scale
* Smokers
* BMI lower than 18.5 or equivalent or higher than 30
* Subjects who had any disease,
* Blood test, urinalysis, physical examination or electrocardiogram showing disorders with clinical relevance
* Subjects receiving treatment for anything apart from contraceptives.
* Gluten, lactose intolerance, vegetarian or vegan subjects for bioequivalence subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-07-09 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Carmen Simón López, RN, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Leticia Carmen Simón López, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The plan is all individual participant data (IPD) that underlie results in a publication. Also, if any volunteer ask for her/his results specifically, a report will be provided.
Supporting Information: Study Protocol, CSR
Time Frame: A Clinical STudy Report is already available for Ethics Committee of La PRINCESA Hospital. Moreover, an original article of the results of the study is being prepared.
Access Criteria: Available as majority as possible.

REFERENCES:
- [Background] de la Torre-Montero JC, Montealegre-Sanz M, Faraldo-Cabana A, Oliva-Pellicer B, Garcia-Real I, Fenwick M, Marcos Caceres E, Rivas-Eguia B, Vila-Borrajo C, Valles-Andres J, Alonso-Gordoa T, Garcia-Carrion C, Diaz-Rubio Garcia E, Beneit-Montesinos JV. Venous International Assessment, VIA scale, validated classification procedure for the peripheral venous system. J Vasc Access. 2014 Jan-Feb;15(1):45-50. doi: 10.5301/jva.5000173. Epub 2013 Sep 4. PMID 24043322
- [Background] Eilers S, Bach DQ, Gaber R, Blatt H, Guevara Y, Nitsche K, Kundu RV, Robinson JK. Accuracy of self-report in assessing Fitzpatrick skin phototypes I through VI. JAMA Dermatol. 2013 Nov;149(11):1289-94. doi: 10.1001/jamadermatol.2013.6101. PMID 24048361
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Fink RM, Hjort E, Wenger B, Cook PF, Cunningham M, Orf A, Pare W, Zwink J. The impact of dry versus moist heat on peripheral IV catheter insertion in a hematology-oncology outpatient population. Oncol Nurs Forum. 2009 Jul;36(4):E198-204. doi: 10.1188/09.ONF.E198-E204. PMID 19581223
- [Background] Yamagami Y, Tomita K, Tsujimoto T, Inoue T. Tourniquet application after local forearm warming to improve venodilation for peripheral intravenous cannulation in young and middle-aged adults: A single-blind prospective randomized controlled trial. Int J Nurs Stud. 2017 Jul;72:1-7. doi: 10.1016/j.ijnurstu.2017.03.009. Epub 2017 Mar 27. PMID 28410510
- [Background] Lima-Oliveira G, Lippi G, Salvagno GL, Montagnana M, Picheth G, Guidi GC. Impact of the phlebotomy training based on CLSI/NCCLS H03-a6 - procedures for the collection of diagnostic blood specimens by venipuncture. Biochem Med (Zagreb). 2012;22(3):342-51. doi: 10.11613/bm.2012.036. PMID 23092065
- [Background] Shah JS, Soon PS, Marsh DJ. Comparison of Methodologies to Detect Low Levels of Hemolysis in Serum for Accurate Assessment of Serum microRNAs. PLoS One. 2016 Apr 7;11(4):e0153200. doi: 10.1371/journal.pone.0153200. eCollection 2016. PMID 27054342
- [Derived] Simon-Lopez LC, Ortuno-Soriano I, Luengo-Gonzalez R, Posada-Moreno P, Zaragoza-Garcia I, Sanchez-Gomez R. Proposal and Strategy for Nursing-Led Research: Protocol for an Unfunded Clinical Trial. JMIR Res Protoc. 2025 Feb 10;14:e56062. doi: 10.2196/56062. PMID 39927682

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 63 individuals signed informed consent form, but one of them did not meet all the inclusion criteria. Then 62 participants were included in the study.
Groups:
- Current Clinical Practice First, Washout, Then Dry Heat: First (day 1): The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week)
  Second (1 day): Dry heat: The application is made with two sacks of carob seeds during 7 minutes. The sacks are placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power.
- Current Clinical Practice First, Washout, Then High Pressure: First (day 1):The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week)
  Second (1 day): High pressure: It will be carried out with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand (QUIRUMED) with European Conformity (CE) marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
- Current Clinical Practice First, Washout, Then Combination: First (day 1): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week)
  Second (1 day): Combination of dry heat and high pressure: as described in dry heat application, and after 7 minutes, high pressure was applied as described for high pressure intervention.
- Dry Heat First, Washout, Then Current Clinical Practice: First ( day 1): Dry heat: The application is made with two sacks of carob seeds during 7 minutes. The sacks are placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power.
  Washout (1 week)
  Second (day 1): The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
- High Pressure First, Washout, Then Current Clinical Practice: First (day 1): High pressure: It will be carried out with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand (QUIRUMED) with European Conformity (CE) marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
  Washout (1 week)
  Second (8 day 1):The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
- Combination First, Washout, Then Current Clinical Practice: First (day 1): Combination of dry heat and high pressure: as described in dry heat application, and after 7 minutes, high pressure was applied as described for high pressure intervention.
  Washout (1 week)
  Second (day 1): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
Period: Overall Study
Arm/Group | Current Clinical Practice First, Washout, Then Dry Heat | Current Clinical Practice First, Washout, Then High Pressure | Current Clinical Practice First, Washout, Then Combination | Dry Heat First, Washout, Then Current Clinical Practice | High Pressure First, Washout, Then Current Clinical Practice | Combination First, Washout, Then Current Clinical Practice
Started | 10 | 11 | 9 | 11 | 10 | 11
Completed | 10 | 8 | 9 | 11 | 10 | 11
Not Completed | 0 | 3 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Current Clinical Practice First, Washout, Then Dry Heat: First (day 1):The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week)
  Second (1 day). Dry heat: The application is made with two sacks of carob seeds during 7 minutes. The sacks are placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power.
- Current Clinical Practice First, Washout, Then High Pressure: First (1 day): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week) .
  Second (1 day): High pressure: It will be carried out with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand (QUIRUMED) with European Conformity (CE) marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
- Current Clinical Practice First, Washout, Then Combination: First (day 1):The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
  Washout (1 week)
  Second (1 day): Combination of dry heat and high pressure: as described in dry heat application, and after 7 minutes, high pressure was applied as described for high pressure intervention.
- Dry Heat First, Washout, Then Current Clinical Practice: First (1 day). Dry heat: The application is made with two sacks of carob seeds during 7 minutes. The sacks are placed on antebrachial anatomical zone, together, and previously heated in the microwave for 0.30 seconds at 850 W of power.
  Washout (1 week)
  Second (day 1):The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
- High Pressure First, Washout, Then Current Clinical Practice: First (1 day): High pressure: It will be carried out with the use of the manual aneroid sphygmomanometer fixed at 100 millimeters of mercury. Brand (QUIRUMED) with European Conformity (CE) marking 0197. A pressure lower than the systolic blood pressure, and in each subject will be monitored the radial pulse.
  Washout (1 week)
  First (1 day): The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
- Combination First, Washout, Then Current Clinical Practice: First (1 day): Combination of dry heat and high pressure: as described in dry heat application, and after 7 minutes, high pressure was applied as described for high pressure intervention.
  Washout (1 week)
  Second (day 1):The standardized and approved CLSI GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
- Total: Total of all reporting groups
Arm/Group | Current Clinical Practice First, Washout, Then Dry Heat | Current Clinical Practice First, Washout, Then High Pressure | Current Clinical Practice First, Washout, Then Combination | Dry Heat First, Washout, Then Current Clinical Practice | High Pressure First, Washout, Then Current Clinical Practice | Combination First, Washout, Then Current Clinical Practice | Total
Number analyzed (Participants) | 10 | 08 | 09 | 11 | 10 | 11 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.33 (3.72) | 30.00 (8.22) | 26.78 (7.80) | 27.36 (3.80) | 26.30 (4.71) | 25.45 (6.91) | 26.72 (5.881)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 4 | 9 | 7 | 7 | 39
  Male | 2 | 4 | 5 | 2 | 3 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 2 | 4 | 3 | 5 | 21
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 5 | 5 | 7 | 7 | 7 | 6 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Grade of Venous International Assessment (VIA) scale [Count of Participants; unit: Participants] — Vein perception in VIA scale was considered as the self-reported visual observation or palpation of a venous pathway.
  Subjects were graded using the current clinical practice vein stagnation with an elastic compressor application (Unidix®).
  Five grades considering the numbers of points of optimal puncture visible and tangible, in one of the dorsal veins of the hand, forearm cephalic and/or basilic.
  Grade I: At least six. Grade II: At least four. Grade III: At least three. Grade IV: At least one. Grade V: None.
  Therefore, the best grade is I, and the worst grade is V.
  Participants
    Grade II | 2 | 3 | 4 | 2 | 1 | 3 | 15
    Grade III | 2 | 3 | 4 | 4 | 1 | 6 | 20
    Grade IV | 6 | 2 | 1 | 4 | 8 | 2 | 23
    Grade V | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Venous Catheterization at the First Attempt
Description: Number of participants with successful venous catheterization at the first attempt (effectiveness)
Time Frame: From 1-5 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Combination: Combination of dry heat and high pressure: The application is made with two sacks of carob seeds during 7 minutes, then application of high pressure as described is carried out.
- Current Clinical Practice: The standardized and approved Clinical and Laboratory Standards Institute (CLSI) GP41-A6 venipuncture guide has been established for clinical current practice so far. According to vein cannulation procedure CLSI GP41-A6, an elastic compressor will be applied (Synthetic rubber-latex compressor tape, UNIDIX®, Madrid, Spain) provided by the hospital.
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
Participants | 21 | 18 | 19 | 28
Statistical Analysis 1: Comparison: Dry Heat vs Current Clinical Practice; Test type: Superiority; p = 0.001, McNemar; Odds Ratio (OR) = 2.57, 95% CI 2-sided [2.34 to 2.79]
Statistical Analysis 2: Comparison: High Pressure vs Current Clinical Practice; Test type: Superiority; p = 0.002, McNemar; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.70 to 2.13]
Statistical Analysis 3: Comparison: Combination vs Current Clinical Practice; Test type: Superiority; p = 0.004, McNemar; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.87 to 1.92]

2. Secondary Outcome: Number of the Grade of Venous International Assessment (VIA) Scale After Application of Intervention
Description: Vein perception in VIA scale was considered as the self-reported visual observation or palpation of a venous pathway.
  Subjects were graded using the current clinical practice vein stagnation with an elastic compressor application (Unidix®).
  Five grades considering the numbers of points of optimal puncture visible and tangible, in one of the dorsal veins of the hand, forearm cephalic and/or basilic.
  Grade I: At least six. Grade II: At least four. Grade III: At least three. Grade IV: At least one. Grade V: None.
  Therefore, the best grade is I, and the worst grade is V. Higher scores mean a worse outcome.
Time Frame: up to ten minutes after application of intervention
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
units on a scale | 2 [1 to 4] | 2 [1 to 4] | 1 [1 to 3] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Dry Heat vs Current Clinical Practice; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney); Median Difference (Net) = -4.179
Statistical Analysis 2: Comparison: High Pressure vs Current Clinical Practice; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney); Median Difference (Net) = -3.619
Statistical Analysis 3: Comparison: Combination vs Current Clinical Practice; Test type: Superiority; p = 0.000, Wilcoxon (Mann-Whitney); Median Difference (Net) = -4.099

3. Secondary Outcome: Number of the Grade in Visual Analogue Scale (VAS) for Pain After Intervention
Description: Visual Analogue Scale (VAS) in pain was measured by integer number. Pain was self-expressed by participants, in a range from 0 to 10.
  10: was considered the worst pain experienced 0: no pain perceived.
  The entire range was 0, 1, 2, 3, 4, 5 , 6, 7, 8, 9, 10.
  Therefore, higher scores mean a worse outcome.
Time Frame: up to 2 hours after application of intervention
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
units on a scale | 3 [0 to 7] | 2 [0 to 6] | 2.5 [0 to 8] | 3 [0 to 8]
Statistical Analysis 1: Comparison: Dry Heat vs Current Clinical Practice; Test type: Superiority; p = 0.863, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.073 — Estimated value corresponds with the number of negative changes, which implies participants with decrease in VAS score
Statistical Analysis 2: Comparison: High Pressure vs Current Clinical Practice; Test type: Superiority; p = 0.205, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.267 — Estimated value corresponds with the number of negative changes, which implies participants with decrease in VAS score
Statistical Analysis 3: Comparison: Combination vs Current Clinical Practice; Test type: Superiority; p = 0.391, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.858 — Estimated value corresponds with the number of negative changes, which implies participants with decrease in VAS score

4. Secondary Outcome: Number of Participants in Each Type of Skin Standardized According to Fitzpatrick Scale
Description: Number of participants in each type of skin standardized according to Fitzpatrick scale. Fitzpatrick scale is the UNABBREVIATED scale that indicates different types of skin described as "phototypes". The individuals were graded clinically by sel-expressed by participants in the area of the forearm not exposed to the sun.
  In a range of six phototypes, where phototype I corresponds with the minimum and phototype VI the maximum.
  Phototype I: Ivory white, burns easily, never tans. Phototype II: White, burns easily, tans minimally with difficulty. Phototype III: White, burns moderately, tans moderately and uniformly Phototype IV: Beige-olive, lightly tanned, burns minimally, tans moderately and easily.
  Phototype V: Rarely burns, tans profusely. Phototype VI: Dark brown or black, never burns, tans profusely.
  Phototype I was considered more risky outcome for expected adverse events in skin. None was considered better or worse outcome.
Time Frame: up to 2 hours after application of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
Participants
  Phototype I | 1 | 1 | 0 | 2
  Phototype II | 2 | 2 | 1 | 5
  Phototype III | 9 | 6 | 8 | 23
  Phototype IV | 7 | 8 | 8 | 23
  Phototype V | 1 | 1 | 3 | 5
  Phototype VI | 1 | 0 | 0 | 1

5. Secondary Outcome: Level of Hemolysis in Absorbance Units
Description: Detection level of absorbance values of hemolysis in plasma samples. The units of absorbance are dimensionless. The hemolysis in plasma is analyzed by spectrophotometry method, using a NanoDrop® 2000 Spectrophotometer device (Thermo Fisher Scientific Inc., Wilmington, United States of America).
  The following equation was used to correct lipemia: (A414-A385) +0.16xA385. Additionally, a baseline correction factor at 750 nanometer wavelength was applied. Therefore, absorbance were measured at 414 nanometer, 385 nanometer and 750 nanometer.
  Higher values represent a worse outcome: higher value mean higher hemolysis in a blood sample.
  Therefore, lower values, near to zero are better outcomes that mean low hemolysis in blood sample.
Time Frame: up to 9 days after first intervention completion
Measure: Median (Full Range); unit: Absorbance units
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
Absorbance units | 0.08 [0.02 to 0.25] | 0.08 [0.06 to 0.60] | 0.14 [0.05 to 0.45] | 0.07 [0.00 to 1.17]
Statistical Analysis 1: Comparison: Dry Heat vs Current Clinical Practice; Test type: Superiority; p = 0.502, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.672 — Estimated value corresponds with the absorbance comparing hemolysis in blood samples performed by clinical practice against to the corresponding intervention
Statistical Analysis 2: Comparison: High Pressure vs Current Clinical Practice; Test type: Superiority; p = 0.744, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.327 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Combination vs Current Clinical Practice; Test type: Superiority; p = 0.059, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.885 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of adverse events by visual inspection.
Time Frame: During the study completion,. an average of 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
Number analyzed (Participants) | 21 | 18 | 20 | 59
Participants | 7 | 1 | 6 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study completion, an average of 30 days.
Description: Because in this clinical trial using dry heat and high pressure were only expected local erythema and transient paresthesia as adverse events. The treatment for those adverse events, if applicable, were not consider a requirement of medical or surgical intervention. A supervision (for local erythema) and release the pressure (for transient paresthesia) were considered sufficient as treatment.
Arm/Group | Dry Heat | High Pressure | Combination | Current Clinical Practice
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/20 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/20 | 0/59
Other Adverse Events (participants affected / at risk) | 7/21 | 1/21 | 6/20 | 0/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dry Heat (N=21) | High Pressure (N=21) | Combination (N=20) | Current Clinical Practice (N=59)
Local erythema (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 6 (6) | 0 (0) — superficial reddening of the skin, usually in patches, as a result of injury or irritation causing dilatation of the blood capillaries.
Transient paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — an abnormal sensation, typically tingling or pricking ('pins and needles'), caused chiefly by pressure on or damage to peripheral nerves.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04027218/Prot_SAP_ICF_001.pdf